CLINICAL TRIAL: NCT06844643
Title: The Disease Progression of Chinese Axial Spondyloarthritis in a Real-word Cohort Study
Acronym: DPCASPA
Status: Recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Weiping Kong, Professor, China-Japan Friendship Hospital
Other Study IDs: 2023-NHLHCRF-YYPPLC-TJ-02
Record Dates: First submitted 2025-02-08; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Axial Spondyloarthritis; Ankylosing Spondylitis (AS)
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
An observational, ambispective cohort to learn about the disease progression of axial spondyloarthritis (axSpA) according to the changes from baseline in measures of disease activity, function, and imaging.

DETAILED DESCRIPTION:
This is an observational cohort study of Chinese patients (≥18 years of age) diagnosed with axSpA. Patients are followed at 4-6 month intervals. Data will be collected at baseline and at every follow-up time points. Primary outcomes are the structural damage measured with imaging(Conventional radiography, low-dose CT and MRI) and the disease activity measured with the Ankylosing Spondylitis Disease Activity Scale (ASDAS) and the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI). Secondary outcomes are inflammatory markers, Bath ankylosing spondylitis functional index (BASFI) and Bath ankylosing spondylitis metrology index (BASMI).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older and diagnosed with the Assessment of Spondyloarthritis International Society axial spondyloarthritis criteria.

Exclusion Criteria:

* Patients with serious disease in cardiovascular, kidney and blood and endocrine system; history of schizophrenia or epilepsy; pregnant or in lactation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with axial spondyloarthritis
Sampling Method: Non-Probability Sample
Enrollment: 2250 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
ASDAS-CRP | From enrollment to 16 weeks, 28 weeks, 1 year; after 1year on a an average of 6 months until study completion.
ASDAS-ESR | From enrollment to 16 weeks, 28 weeks, 1 year; after 1year on a an average of 6 months until study completion.
BASDAI | From enrollment to 16 weeks, 28 weeks, 1 year; after 1year on a an average of 6 months until study completion.
Modified stoke ankylosing spondylitis spinal score (mSASSS) | 2-year interval
  The mSASSS is a valid and widely used method for assessing radiographic progression in AS, correlating with worsening measures of disease signs and symptoms, spinal mobility and physical function.
The Spondyloarthritis Research Consortium of Canada (SPARCC) scoring system. | From enrollment to 16 weeks，1 year; after 1year on a an average of 6 months until study completion.
  The Spondyloarthritis Research Consortium of Canada (SPARCC) developers have created the SPARCC MRI scoring methods to assess inflammatory activity in patients with SpA.

SECONDARY OUTCOMES:
BASFI | From enrollment to 16 weeks, 28 weeks, 1 year; after 1year on a an average of 6 months until study completion.
BASMI | From enrollment to 16 weeks, 28 weeks, 1 year; after 1year on a an average of 6 months until study completion.

OTHER OUTCOMES:
CT Syndesmophyte Score | 2-year interval
  The CT Syndesmophyte Score (CTSS) was developed for the assessment of syndesmophytes on LDCT images.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No